CLINICAL TRIAL: NCT05968651
Title: Social Safety Learning in the Brain Oxytocin System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Angela Fang, Assistant Professor, Department of Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00013670
Record Dates: First submitted 2023-07-10; First posted 2023-08-01 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Social Phobia
Keywords: Social Phobia; Social Anxiety Disorder; Social Safety Learning; Intranasal Oxytocin
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical (Experimental): This group consists of individuals with at least moderate symptoms of social anxiety disorder. This group will receive either an oxytocin or placebo administration (blind randomization).
  Interventions: Drug: Oxytocin nasal spray
- Controls (Placebo Comparator): This group consists of a healthy sample of individuals (no lifetime diagnoses of mania or psychotic disorders). This group will receive either an oxytocin or placebo administration (blind randomization).
  Interventions: Drug: Oxytocin nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — Single acute administration of 24 international units (IU) oxytocin

SUMMARY:
The investigators are conducting this research study to examine whether oxytocin enhances social safety learning (learning safety through the experience of another individual) in people with social anxiety disorder (SAD) compared to healthy volunteers. Oxytocin is a hormone that can also act as a chemical messenger in the brain. Oxytocin plays a role in a number of functions, including responding to fear and social interactions. In this study, the investigators would like to compare the effects of oxytocin and placebo nasal sprays in adults with SAD and healthy adults. This research study will compare an oxytocin nasal spray to a placebo nasal spray. About 120 people will take part in this research study, all at the University of Washington (UW).

DETAILED DESCRIPTION:
The goal of the current study is to examine the potential role of oxytocin in enhancing social learning in SAD. The investigators' primary hypothesis is that vicarious extinction learning will contribute to safety learning and that oxytocin will potentiate vicarious extinction learning in patients with SAD, compared to healthy controls (HC). The investigators will directly test the effect of intranasal oxytocin and matching placebo on the brain mechanisms underlying vicarious extinction learning using a novel task. 60 adults with SAD and 60 healthy control participants will perform a task that involves three phases: (i) a standard social fear acquisition procedure while in a mock scanner, followed by (ii) a vicarious extinction and (iii) fear reinstatement test procedure, while being scanned during functional magnetic resonance imaging (fMRI). Participants will receive oxytocin or placebo prior to the extinction phase. The investigators will also measure skin conductance responses as an index of learning in each phase.

ELIGIBILITY:
Inclusion Criteria:

For Clinical Sample

* Men and women age 18-45
* Women must be having regular menstrual cycles and not be taking oral contraception
* Primary diagnosis of social anxiety disorder

For Healthy Sample

* Men and women age 18-45
* Women must be having regular menstrual cycles and not be taking oral contraception
* No current or lifetime history of psychiatric, neurological, or medical disorders

Exclusion Criteria:

For All Groups

* Pregnancy or breastfeeding
* Positive urine drug screening test result
* History of nasal pathology
* Current use of any psychotropic medication or steroids
* Active substance use disorder within the past 6 months
* History of serious medical illnesses or untreated endocrine diseases
* History of head injury, neurological disorder, or neurosurgical procedure
* Positive magnetic resonance (MR) screen

For Clinical Sample

* Lifetime diagnoses of mania or psychotic disorder based on the Diagnostic and Statistical Manual (DSM- 5th ed)
* Acute suicidal ideation

For Healthy Sample

* Lifetime DSM-5 diagnosis of any medical, neurological, or psychiatric illness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
neural responses (e.g., regional brain activation in the ventromedial prefrontal cortex (vmPFC) to vicariously extinguished cue versus vicariously reinforced cue during reinstatement | immediately after the intervention
  vmPFC blood oxygen level dependent (BOLD) responses for non-reinforced conditioned stimulus (CS-) versus reinforced conditioned stimulus (CS+)

SECONDARY OUTCOMES:
skin conductance responses (SCR) to vicariously extinguished cue versus vicariously reinforced cue during reinstatement | immediately after the intervention
  mean SCR for CS- versus CS+

CONTACTS AND LOCATIONS:
Overall Officials: Angela Fang, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No